CLINICAL TRIAL: NCT05881213
Title: A Randomized, Open-label, Single-dose, Two-way Crossover Clinical Trial to Investigate the Pharmacokinetics and Safety After Oral Administration of CKD-378 and Co-administration of D745, D150, D029 in Healthy Adults
Brief Title: Clinical Trial to Investigate the Pharmacokinetics and Safety After Oral Administration of CKD-378 and Co-administration of D745, D150, D029 in Healthy Adults
Acronym: CKD-378
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: A129_02BE2227
Record Dates: First submitted 2023-05-18; First posted 2023-05-31 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-05

CONDITIONS: Type II Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence 1 (Experimental): * Period 1: D745, D150, D029 - A single oral dose of 3tablets under food intake condition
  * Period 2: CKD-378 (low-dose) - A single oral dose of 1tablet under food intake condition
  Interventions: Drug: CKD-378 (low-dose)
- Sequence 2 (Experimental): * Period 1: CKD-378 (low-dose) - A single oral dose of 1tablet under food intake condition
  * Period 2: D745, D150, D029 - A single oral dose of 3tablets under food intake condition
  Interventions: Drug: CKD-378 (low-dose)

INTERVENTIONS:
Drug: CKD-378 (low-dose) — Quaque day (QD), PO

SUMMARY:
A clinical trial to compare and evaluate the safety and pharmacokinetics of CKD-378

DETAILED DESCRIPTION:
A Randomized, Open-label, Single-dose, Two-way Crossover Clinical Trial to Investigate the Pharmacokinetics and Safety after Oral Administration of CKD-378 and Co-administration of D745, D150, D029 in Healthy Adults

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults aged between 19 and 55 years at screening.
2. Those whose body weight 55 kg or over for men and 50 kg or over for women.
3. Those with body mass index (BMI) was more than 18.5 kg/m2 and less than 27.0 kg/m2.

   ※ BMI (kg/m2) = body weight (kg)/ [height (m)]2
4. If women, those who met any one of the following criteria.

   * Menopause (no natural menstruation for at least 2 years)
   * Surgical infertility (hysterectomy or bilateral oophorectomy, tubal ligation, or infertility by other methods)
5. Male subjects with female sexual partners of childbearing potential must agree to use methods of birth control (using condom) and not donate sperm during the study and for up to 28 days after the last administration of the IP (unless the male subjects or their female partners are infertile).
6. Subjects who have voluntarily given written informed consent to participate in the study and comply with all study requirements after getting a detailed explanation and full understanding of the study.

Exclusion Criteria:

1. Subjects with history or current conditions of clinically significant disease, including hepatobiliary (e.g., severe hepatic dysfunction, etc.), renal (e.g., severe renal insufficiency, etc.), nervous, immune, respiratory (e.g., bronchial asthma) urinary, gastrointestinal, endocrine (e.g., patients with diabetic ketoacidosis, diabetic coma and pre-coma, and type 1 diabetes mellitus, etc.), hemato-oncology, or cardiovascular (e.g., heart failure, etc.) or psychiatric disorders.
2. Subjects who are susceptible to dehydration due to inadequate oral intake or who have clinically significant dehydration.
3. Subjects who underwent a test using intravenous administration of radioiodine contrast media (e.g., intravenous urography, venous cholangiography, angiography, or computed tomography using a contrast medium) within 48 hours prior to the first IP administration.
4. Subjects with a history or current conditions of serious urinary tract infection.
5. Subjects with genetic problems such as galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption.
6. Subjects with a history of gastrointestinal disorders (e.g., Crohn's disease, ulcerative colitis, etc.) or surgery (except simple appendectomy or hernia surgery) that may affect the absorption of IP.
7. Subjects with a history of clinically significant hypersensitivity to drugs, including components of the IPs (empagliflozin or metformin) or additives.
8. Subjects who were deemed unfit for participation in this study based on the following findings in the screening tests performed within 28 days before the first IP administration.

   * Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) values > 1.25 times the upper limit of normal range.
   * Estimated glomerular filtration rate (eGFR) < 60 mL/min/1.73 m2 when calculated with the modification of diet in renal disease (MDRD) formula.
   * Positive result for hepatitis B, hepatitis C, human immunodeficiency virus (HIV), or syphilis infection test.
   * Systolic blood pressure > 150 mmHg or <90 mmHg, or diastolic blood pressure > 100 mmHg or <50 mmHg which is measured in sitting position after resting for more than 5 minutes.
9. Subjects with a history of drug abuse within a year prior to screening or positive results in urine drug screening tests.
10. Women who are pregnant or breast-feeding.
11. Subjects who took the following drugs, excluding the topical agents without significant systemic absorption, within the predefined period the investigator judges they could affect the results of the study or compromise the safety of the subject.

    * Any prescription drugs and herbal medicines within 14 days before the first IP administration.
    * Any over-the-counter drugs including health care foods or vitamins within 7 days before the first IP administration
    * Any drugs administered by depot injection or other implantation into the body within 30 days before the first IP administration
12. Subjects who took any drugs that induce or inhibit drug metabolizing enzymes, such as barbital drugs, within 30 days before the first IP administration.
13. Subjects with excessive smoking (>10 cigarette/day), caffeine intake (caffeine:>5 cups/day), or drinking (alcohol: >210 g/week) or who cannot stop from smoking, caffeine intake, and drinking during the hospitalization period.
14. Subjects who have consumed foods containing grapefruit within 7 days prior to the first IP administration or cannot stop consuming foods containing grapefruit during the study.
15. Subjects who were administered any other IPs by participating in other clinical trials within 180 days before the first IP administration (in the case of biological agent, taking account of its half-life, this period can be extended).
16. Subjects who donated whole blood within 60 days or blood components for apheresis within 30 days before the first IP administration.
17. Subjects who received blood transfusion within 30 days before the first IP administration.
18. Subjects judged by the investigators unsuitable for participating in the study based on any other reasons.

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-06-28 (Actual); Study Completion 2023-07-10 (Actual)

PRIMARY OUTCOMES:
area under the curve (AUC)t of CKD-378 | Pre-dose(0 hour) to 48 hours
  Area under the concentration-time curve time zero to time
Cmax of CKD-378 | Pre-dose(0 hour) to 48 hours
  Maximum plasma concentration of the drug

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No